CLINICAL TRIAL: NCT03744546
Title: Expanded Access to ABBV-8E12
Status: No longer available | Type: Expanded Access
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: C19-364; C19-921 (Other Grant/Funding Number: AbbVie)
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Primary Tauopathy Corticobasal Degeneration Syndrome (CBD)
Keywords: Expanded Access, Pre-approval Access, Compassionate Use, Special Access Program, Named Patient Basis, Special Access Scheme.
MeSH Terms: interventions — tilavonemab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: ABBV-8E12 — Solution for infusion

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to ABBV-8E12 prior to approval by the local regulatory agency. Availability will depend on territory eligibility. Participating sites will be added as they apply for and are approved for the EAP. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

Min Age: 40 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie